CLINICAL TRIAL: NCT06070194
Title: Cardiovascular Risk and Circadian Misalignment in Short Sleepers - Role of Extended Eating Period
Acronym: CRISP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Prachi Singh, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PBRC 2023-025; R01HL166306 (NIH)
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sleep Deprivation
Keywords: eating duration; short sleep duration; time-restricted eating; blood pressure; insulin resistance
MeSH Terms: conditions — Sleep Deprivation; Intermittent Fasting; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (TRE) (Experimental): Subjects randomized to this arm will be asked to follow an 8h eating duration/day for 4 weeks.
  Interventions: Behavioral: Time restricted eating (TRE)
- Habitual eating duration (No Intervention): Subjects randomized to this arm will be asked to continue habitual eating duration of >14h/day for 4 weeks.

INTERVENTIONS:
Behavioral: Time restricted eating (TRE) — Subjects randomized to this arm will be asked to follow an 8h eating duration/day for 4 weeks. Participants will be asked to continue habitual sleep patterns.
  Arms: Time restricted eating (TRE)

SUMMARY:
Short sleep duration confers high cardiovascular and metabolic risk, but lifestyle factors and molecular mechanisms that contribute to increased blood pressure and poor glucose control during short sleep are not completely understood. Habitual short sleepers are constantly eating, the proposed studies will evaluate if this behavior contributes to heightened cardiovascular and metabolic risk. The study will evaluate if restricted eating duration (8 hours/day) could improve cardiovascular and metabolic health in habitual short sleepers.

DETAILED DESCRIPTION:
Short sleep duration is associated with increased cardiovascular and metabolic risk with consequent increased cardiovascular mortality. Increasing sleep duration mitigates the metabolic impairment, but alternate strategies to reduce cardiometabolic risk in habitual short sleepers are lacking. This is especially important when increasing sleep duration is unsuccessful. Unfortunately, the underlying mechanisms through which shortened sleep contributes to metabolic detriments are not completely understood. This hinders the development of alternate strategies for cardiovascular prevention in short sleepers. However, a widespread factor potentially underlying metabolic dysfunction in short sleepers seems to be circadian misalignment (decreased and delayed melatonin secretion) partly resulting from mistimed eating. Importantly, eating behavior may be targeted to improve metabolism in short sleepers. Specifically, limiting the daily eating period as shown by the many recent interventions of time restricted eating (TRE) may potentiate circadian alignment (melatonin rhythms) and improve metabolism in habitual short sleepers.

The goal of the study is to examine the metabolic and circadian effects of eating duration in habitual short sleepers. The investigators propose a two-group, parallel arm study during which participants will be randomized to either continue with habitual >14h/day (extended) or restricted 8h/day (TRE) eating duration. The overarching hypothesis is that extended eating duration contributes to high blood pressure (BP), insulin resistance (IR), and a decreased and delayed melatonin secretion in habitual short sleepers. Therefore, TRE will reduce BP, IR along with an increased and earlier onset of melatonin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years
* BMI: 25-35 kg/m2
* Habitual sleep duration: ≤6.5 h/night
* Habitual eating period: >14h/day
* Absence of chronic health conditions including hypertension (defined as systolic clinical BP of >140 or diastolic BP of >90 mmHg or use of BP lowering drugs), dyslipidemia (defined as LDL >190mg/dL or Triglycerides >400 mg/dL or use of lipid lowering medications), diabetes (defined as fasting glucose >126 mg/dL and /or HbA1C >6.5%, or use of glucose lowering medication), and cardiovascular disease. However, individuals with prehypertension, and/or prediabetes will be allowed to participate.
* Individuals with seasonal allergies will also be included.
* Women of child-bearing age will be allowed to participate if they agree to use acceptable birth control during the study period.
* Must be able to provide written informed consent.
* Ability to follow the prescribed eating duration and maintain habitual diet, sleep and physical activity.
* Use of certain mediations will be allowed including birth control, second generation antihistamines, antacids, acne-related ointments etc.

Exclusion Criteria:

* Irregular sleep habits / night shift / rotating shift work in past 1 month.
* Frequent travel related jet lag.
* Pregnant/ breast-feeding/ history of irregular menstrual cycles.
* Sleep disorders such as insomnia (defined as Insomnia Severity Index score ≥15), and sleep apnea (overnight oximetry defined oxygen desaturation index of >10 events/h of sleep).
* Presence of excessive daytime sleepiness (defined as Epworth Sleepiness Scale score >10).
* Recent changes in body weight (≥5%) within 3 months.
* Uncontrolled depression and /or anxiety, history of psychosis or bipolar disorder.
* Uncontrolled depression and/or depression is defined as PHQ-9 score of ≥15 or a positive response for suicidal thoughts (Q9 of the PHQ-9 - any response other than not at all).
* Any medication or condition that, in the opinion of the medical investigator, could interfere with the study outcomes or put the subject at risk by participating in the study.
* Blood or plasma donation during the past 2 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in 24h mean arterial blood pressure (MAP) | Baseline to 4 weeks
  Change in 24h MAP from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.
Change in insulin resistance | Baseline to 4 weeks
  Change in insulin resistance from pre-intervention to end-intervention. Insulin resistance will be determined by standard 3h mixed meal tolerance test and calculated as ratio of incremental area under the curve values for insulin and glucose. Difference between habitual eating period and TRE will be evaluated.

SECONDARY OUTCOMES:
Change in 24h systolic blood pressure (SBP) | Baseline to 4 weeks
  Change in 24h SBP from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.
Change in postprandial glycemic excursion | Baseline to 4 weeks
  Change in postprandial glycemic excursion from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.

OTHER OUTCOMES:
Change in clock time for dim light melatonin onset | Baseline to 4 weeks
  Change in clock time for dim light melatonin onset from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.
Change in clock time for dim light melatonin offset | Baseline to 4 weeks
  Change in clock time for dim light melatonin offset from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.
Change in melatonin area under the curve (AUC) | Baseline to 4 weeks
  Change in AUC from melatonin onset to offset from pre-intervention to end-intervention. Difference between habitual eating period and TRE will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Singh, PhD, Principal Investigator — Pennington Biomedical Research Institute
Locations (1):
- Recruiting core Pennington, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No